CLINICAL TRIAL: NCT03180736
Title: A Phase 3 Study Comparing Pomalidomide and Dexamethasone With or Without Daratumumab in Subjects With RRMM Who Have Received at Least One Prior Line of Therapy With Both Lenalidomide and a Proteasome Inhibitor.
Brief Title: Comparison of Pom and Dex in Subjects With RRMM Previously Treated With Len and a PI Dara/Pom/Dex vs Pom/Dex
Acronym: EMN14
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMN14/54767414MMY3013
Record Dates: First submitted 2017-05-30; First posted 2017-06-08 (Actual); Results first posted 2022-05-11 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; darlin protein, Dictyostelium; pomalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Intervention Model: Parallel Assignment Masking: Open Label Primary Purpose: Treatment
Who Masked: Participant
Masking Description: Masking: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daratumumab+Pomalidomide+Dexamethasone (Experimental): Daratumumab at a dose of 16 mg/kg administered as an IV infusion (Dara IV) or 1800 mg subcutaneously (Dara SC) at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Pomalidomide 4 mg orally (PO) on Days 1 through 21 of each 28-day cycle Dexamethasone 40 mg (20 mg for patients ≥75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle
  Interventions: Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone
- Pomalidomide + Dexamethasone (Active Comparator): Pomalidomide 4 mg orally (PO) on Days 1 through 21 of each 28-day cycle Dexamethasone 40 mg (20 mg for patients ≥75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be given at a dose of 16 mg/kg administered as an IV infusion (Dara IV) or 1800 mg subcutaneously (Dara SC) at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, then every 4 weeks (Q4W) thereafter. Subjects will receive pre-infusion medications before infusions to mitigate potential IRRs.
  Other Names: Dara
  Arms: Daratumumab+Pomalidomide+Dexamethasone
Drug: Pomalidomide — Pomalidomide will be administered at full dose of 4 mg orally (PO) on Days 1 through 21 of each 28-day cycle.
  Other Names: Pom
Drug: Dexamethasone — Dexamethasone will be administered at a dose of 40 mg (20 mg for patients ≥75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
  Other Names: Dex

SUMMARY:
The purpose of this study is to evaluate the effects of the addition of daratumumab to pomalidomide and dexamethasone in terms of progression-free survival in subjects with relapsed or refractory Multiple Myeloma.

DETAILED DESCRIPTION:
This is a multicenter, Phase 3, randomized, open-label study comparing daratumumab, pomalidomide and low-dose dexamethasone (DaraPomDex) with pomalidomide and low-dose dexamethasone (PomDex) in subjects with relapsed or refractory Multiple Myeloma who have received at least 1 prior treatment regimen with both lenalidomide and a proteasome inhibitor and have demonstrated disease progression. Subjects will be randomized in a 1:1 ratio to receive either DaraPomDex or PomDex. The original design of this study was to treat subjects with daratumumab for intravenous (IV) infusion (Dara IV); however, as of Amendment 1, all new subjects will be dosed subcutaneously with daratumumab co-formulated with recombinant human hyaluronidase rHuPH20 (hereafter referred to as Dara SC). Subjects who already began treatment with Dara IV (ie, prior to Amendment 1) will have the option to switch to Dara SC on Day 1 of any cycle starting with Cycle 3 or later for the remainder of their participation in the study, and they will be counted toward the total of 302 subjects. Subjects will receive treatment until disease progression or unacceptable toxicity. Drug administration and follow-up visits will occur more frequently for early cycles (e.g., weekly or bi-weekly). Disease evaluations will occur every cycle and consist mainly of measurements of myeloma proteins. Subject safety will be assessed throughout the study. The primary endpoint will be progression-free survival (PFS). Study end is anticipated at approximately 5 years after the last subject is randomized.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females at least 18 years of age.
2. Voluntary written informed consent before performance of any study-related procedure.
3. Subject must have measurable disease of MM as defined by the criteria below:

   * IgG multiple myeloma: Serum M protein level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours, or
   * IgA, IgD, IgE, IgM multiple myeloma: Serum M-protein level ≥0.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
   * Light chain multiple myeloma, for subjects without measurable disease in the serum or urine: Serum immunoglobulin free light chain (FLC) ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
4. Subjects must have received prior antimyeloma treatment. The prior treatment must have included both a PI- and lenalidomide-containing regimens. The subject must have had a response (ie, PR or better based on the investigator's determination of response as defined by the modified IMWG criteria) to prior therapy.
5. Subjects must have documented evidence of PD based on the investigator's determination of response as defined by the modified IMWG criteria on or after the last regimen.
6. Subjects who received only 1 line of prior treatment must have demonstrated PD on or within 60 days of completion of the lenalidomide containing regimen (ie, lenalidomide refractory).
7. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤ 2.
8. Willingness and ability to participate in study procedures.
9. For subjects experiencing toxicities resulting from previous therapy, the toxicities must be resolved or stabilized to ≤Grade 1.
10. Any of the following laboratory test results during Screening:

    1. Absolute neutrophil count ≥1.0 × 109/L;
    2. Hemoglobin level ≥7.5 g/dL (≥4.65 mmol/L); (transfusions are not permitted to reach this level);
    3. Platelet count ≥75 × 109/L in subjects in whom <50% of bone marrow nucleated cells are plasma cells and platelet count ≥50 x 109/L in subjects in whom ≥50% of bone marrow nucleated cells are plasma cells;
    4. Alanine aminotransferase (ALT) level ≤2.5 times the upper limit of normal (ULN);
    5. Aspartate aminotransferase (AST) level ≤2.5 x ULN;
    6. Total bilirubin level ≤1.5 x ULN, (except for Gilbert Syndrome: direct bilirubin ≤1.5 × ULN);
    7. Creatinine clearance ≥30 mL/min
    8. Serum calcium corrected for albumin ≤14.0 mg/dL (≤3.5 mmol/L), or free ionized calcium ≤ 6.5 mg/dL (≤1.6 mmol/L).
11. Reproductive Status

    1. Women of childbearing potential (WOCBP) must have 2 negative serum or urine pregnancy tests, one 10-14 days prior to start of study treatment and one 24 hours prior to the start of study treatment. Females are not of reproductive potential if they have been in natural menopause for at least 24 consecutive months, or have had a hysterectomy and/or bilateral oophorectomy.
    2. Women must not be breastfeeding.
    3. WOCBP must agree to follow instructions for methods of contraception for 4 weeks before the start of study treatment, for the duration of study treatment, and for 3 months after cessation of daratumumab or 4 weeks after cessation of pomalidomide, whichever is longer.
    4. Males who are sexually active must always use a latex or synthetic condom during any sexual contact with females of reproductive potential, even if they have undergone a successful vasectomy. They must also agree to follow instructions for methods of contraception for 4 weeks before the start of study treatment, for the duration of study treatment, and for a total of 3 months post-treatment completion.
    5. Male subjects must not donate sperm for up to 90 days post-treatment completion.
    6. Female subject must not donate eggs for up to 90 days post-treatment completion.
    7. Azoospermic males and WOCBP who are not heterosexually active are exempt from contraceptive requirements. However, WOCBP will still undergo pregnancy testing as described in this section.

Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly. Subjects must agree to the use of 2 methods of contraception, with 1 method being highly effective and the other method being additionally effective.

Because of the embryo-fetal risk of pomalidomide, all subjects must adhere to the pomalidomide pregnancy prevention program applicable in their region. Investigators should comply with the local label for pomalidomide for specific details of the program.

Exclusion Criteria:

1. Previous therapy with any anti-CD38 monoclonal antibody.
2. Previous exposure to pomalidomide.
3. Subject has received antimyeloma treatment within 2 weeks or 5 pharmacokinetic half-lives of the treatment, whichever is longer, before the date of randomization. The only exception is emergency use of a short course of corticosteroids (equivalent of dexamethasone 40 mg/day for a maximum of 4 days) for palliative treatment before Cycle 1, Day 1 (C1D1).
4. Previous allogenic stem cell transplant; or autologous stem cell transplantation (ASCT) within 12 weeks before C1D1.
5. History of malignancy (other than MM) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 3 years).
6. Clinical signs of meningeal involvement of MM.
7. Chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
8. Clinically significant cardiac disease, including:

   1. Myocardial infarction within 6 months, before C1D1 or unstable or uncontrolled condition (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV).
   2. Cardiac arrhythmia (Common Terminology Criteria for Adverse Events [CTCAE] Grade 3 or higher) or clinically significant electrocardiogram (ECG) abnormalities.
   3. Electrocardiogram showing a baseline QT interval as corrected QTc >470 msec.
9. Known active hepatitis A, B, or C.
10. Known HIV infection.
11. Gastrointestinal disease that may significantly alter the absorption of pomalidomide.
12. Subject has plasma cell leukemia (>2.0 × 109/L circulating plasma cells by standard differential) or Waldenström's macroglobulinemia or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes) or amyloidosis.
13. Any concurrent medical or psychiatric condition or disease (eg, active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results or that, in the opinion of the investigator, would constitute a hazard for participating in this study.
14. Ongoing ≥ Grade 2 peripheral neuropathy.
15. Subject had ≥Grade 3 rash during prior therapy.
16. Subject has had major surgery within 2 weeks before randomization, or has not fully recovered from an earlier surgery, or has surgery planned during the time the subject is expected to participate in the study or within 2 weeks after the last dose of study drug administration. Note: subjects with planned surgical procedures to be conducted under local anesthesia may participate. Kyphoplasty or vertebroplasty are not considered major surgery.
17. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof, Principal Investigator — Department of Clinical Therapeutics, University of Athens, School of Medicine, Athens, Greece
Locations (40):
- Belgium (4):
  - Antwerpen, Antwerp
  - Brussel, Brussels
  - UZ Gent, Ghent
  - Yvoir, Yvoir
- Czechia (3):
  - Brno, Brno
  - Ostrava, Ostrava
  - Praha 2, Prague
- Denmark (2):
  - Odense, Odense
  - Vejle, Vejle
- Germany (7):
  - Freiburg, Freiburg im Breisgau
  - Hamburg, Hamburg
  - Heidelberg, Heidelberg
  - Kiel, Kiel
  - Schwerin, Schwerin
  - Tübingen, Tübingen
  - Würzburg, Würzburg
- Greece (4):
  - General Hospital of Athens "Evangelismos", Athens
  - University of Athens School of Medicine, Athens
  - General University Hospital of Patras, Pátrai
  - Anticancer Hospital of Thessaloniki "Theageneio", Thessaloniki
- Italy (6):
  - Ancona, Ancona
  - Bologna, Bologna
  - Brescia, Brescia
  - Milano, Milan
  - Roma, Roma
  - Torino, Torino
- Netherlands (2):
  - VU MC, Amsterdam
  - Erasmus MC, Rotterdam
- Belgrade, Belgrade, Serbia
- Spain (6):
  - Badalona, Badalona
  - Barcelona, Barcelona
  - Hospital Quirón Salud Madrid, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Salamanca University Hospital, Salamanca
  - Doctor Peset University Hospital Medical Centre, Valencia
- Turkey (Türkiye) (5):
  - Cebeci, Cebeli
  - Capa, Çapa
  - Gaziantep, Gaziantep
  - Izmir, Izmir
  - Kayseri, Kayseri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dimopoulos MA, Terpos E, Boccadoro M, Delimpasi S, Beksac M, Katodritou E, Moreau P, Baldini L, Symeonidis A, Bila J, Oriol A, Mateos MV, Einsele H, Orfanidis I, Kampfenkel T, Liu W, Wang J, Kosh M, Tran N, Carson R, Sonneveld P. Subcutaneous daratumumab plus pomalidomide and dexamethasone versus pomalidomide and dexamethasone in patients with relapsed or refractory multiple myeloma (APOLLO): extended follow up of an open-label, randomised, multicentre, phase 3 trial. Lancet Haematol. 2023 Oct;10(10):e813-e824. doi: 10.1016/S2352-3026(23)00218-1. PMID 37793772
- [Derived] He J, Berringer H, Heeg B, Ruan H, Kampfenkel T, Dwarakanathan HR, Johnston S, Mendes J, Lam A, Bathija S, Mackay EK. Indirect Treatment Comparison of Daratumumab, Pomalidomide, and Dexamethasone Versus Standard of Care in Patients with Difficult-to-Treat Relapsed/Refractory Multiple Myeloma. Adv Ther. 2022 Sep;39(9):4230-4249. doi: 10.1007/s12325-022-02226-x. Epub 2022 Jul 22. PMID 35876974
- [Derived] Dimopoulos MA, Terpos E, Boccadoro M, Delimpasi S, Beksac M, Katodritou E, Moreau P, Baldini L, Symeonidis A, Bila J, Oriol A, Mateos MV, Einsele H, Orfanidis I, Ahmadi T, Ukropec J, Kampfenkel T, Schecter JM, Qiu Y, Amin H, Vermeulen J, Carson R, Sonneveld P; APOLLO Trial Investigators. Daratumumab plus pomalidomide and dexamethasone versus pomalidomide and dexamethasone alone in previously treated multiple myeloma (APOLLO): an open-label, randomised, phase 3 trial. Lancet Oncol. 2021 Jun;22(6):801-812. doi: 10.1016/S1470-2045(21)00128-5. PMID 34087126

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were randomly allocated to 1 of the 2 arms (Pd or DPd). 7 patients started with daratumumab IV. The study was amended to daratumumab SC formulation. Of those 7 patients, 4 switched to daratumumab SC and 3 discontinued treatment before the study was amended to SC administration. All other daratumumab-treated patients (142 of 149 DPd subjects) received only daratumumab SC. In summary, almost all patients (146 of 149) that were treated in the DPd arm received daratumumab SC.
Groups:
- Daratumumab+Pomalidomide+Dexamethasone: Patients received Daratumumab subcutaneously (fixed dose of 1800 mg) or intravenously (16 mg/kg) weekly for cycles 1-2, every 2 weeks for cycles 3-6, and every 4 weeks thereafter. Pomalidomide was administered at a dose of 4 mg orally every day on days 1 through 21, and dexamethasone at 40 mg (or 20 mg for patients ≥75 years of age) orally weekly, in 28-day cycles..
  Pomalidomide: Pomalidomide will be administered at full dose of 4 mg orally (PO) on Days 1 through 21 of each 28-day cycle.
  Dexamethasone: Dexamethasone will be administered at a dose of 40 mg (20 mg for patients ≥75 years of age) orally, once daily on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
- Pomalidomide + Dexamethasone: Patients received Pomalidomide at a dose of 4 mg orally every day on days 1 through 21, and dexamethasone 40 mg (or 20 mg for patients ≥75 years of age) orally weekly, in 28-day cycles
Period: Overall Study
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Started | 151 | 153
Treated | 149 | 150
Completed | 60 | 33
Not Completed | 91 | 120
Not completed — Adverse Event | 3 | 4
Not completed — Death | 10 | 7
Not completed — Withdrawal by Subject | 5 | 12
Not completed — Lost to Follow-up | 1 | 0
Not completed — Lack of Efficacy | 66 | 87
Not completed — Physician Decision | 4 | 7
Not completed — randomized but not treated | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone | Total
Number analyzed (Participants) | 151 | 153 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (9.57) | 66.5 (9.70) | 66.0 (9.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 71 | 143
  Male | 79 | 82 | 161
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Greece | 53 | 44 | 97
  Netherlands | 5 | 4 | 9
  Turkey | 16 | 24 | 40
  Belgium | 7 | 9 | 16
  Czechia | 6 | 4 | 10
  Denmark | 1 | 1 | 2
  Italy | 19 | 20 | 39
  Serbia | 4 | 5 | 9
  Germany | 8 | 7 | 15
  Spain | 15 | 22 | 37
  Poland | 1 | 1 | 2
  France | 16 | 12 | 28
Stage of Disease (ISS) [Count of Participants; unit: Participants] — The International Staging System (ISS) consists of the following 3 stages; Stage I: serum beta2-microglobulin less than (<) 3.5 milligram per liter (mg/L) and albumin greater than or equal to (≥) 3.5 gram per 100 Milliliter (g/100 mL); Stage II: neither stage I nor stage III; and Stage III: serum beta2-microglobulin greater than or equal to (≥) 5.5 mg/L. Higher stages indicate more severe disease (i.e. worse outcomes).
  Participants
    I | 68 | 69 | 137
    II | 50 | 51 | 101
    III | 33 | 33 | 66
No. of Prior Lines of Therapy [Count of Participants; unit: Participants]
  1 | 16 | 18 | 34
  2-3 | 114 | 113 | 227
  ≥4 | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Progression Free Survival Between Treatment Arms (Daratumumab /Pomalidomide /Dexamethasone vs Pomalidomide / Dexamethasone)
Description: Progression Free Survival (PFS) is defined as the time, in months, from randomization to the date of the first documented disease progression (PD) or death due to any cause, whichever comes first.
  PFS2 is defined as the time, in months, from randomization to the date of the first documented disease progression (PD) or death due to any cause, whichever comes first, after the next line of therapy.
  PD is assessed by the investigator based on the analysis of serum and urine protein electrophoresis (sPEP and uPEP), serum and urine immunofixation (sIFE and uIFE), serum free light chain protein (sFLC),corrected serum calcium assessment, imaging and bone marrow assessments as per modified IMWG guidelines.
Time Frame: PFS is assessed monthly from randomization until PD or death, whichever occurs first (approximately up to 3 years). PFS2 is assessed monthly from randomization until PD or death, whichever occurs first (approximately up to 5 years).
Population: The intent-to-treat (ITT) analysis set includes all participants who were randomly assigned to the pomalidomide, dexamethasone (Pd) or daratumumab, pomalidomide, dexamethasone (DPd) group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
months
  PFS2: number analyzed (Participants) | 88 | 105
  PFS2 | 24.41 [17.05 to 35.71] | 17.58 [13.57 to 21.98]
  Primary Efficacy of PFS | 12.42 [8.34 to 19.32] | 6.93 [5.52 to 9.26]

2. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the proportion of randomized participants who achieved a best response of PR or better using modified IMWG criteria.
Time Frame: Approximately up to 3 years (assessed monthly from randomization until PD).
Population: The intent-to-treat (ITT) population was used for efficacy evaluations (total of 304 randomized subjects, 151 in the Daratumumab/Pomalidomide/Dexamethasone group and 153 in the Pomalidomide/Dexamethasone group).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
percentage of participants | 68.87 [60.84 to 76.15] | 46.41 [38.32 to 54.64]

3. Secondary Outcome: Depth of Response
Description: Depth of response is the analysis of the Minimal Residual Disease (MRD) negativity rate at the sensitivity threshold of 10^-5 for patients who have achieved CR or better and for patients with suspected CR/sCR.
Time Frame: MRD is assessed at the time of suspected CR/sCR and 6, 12, 18, 24, and every 12 months (yearly assessments ±3 months) post CR/sCR in subjects who maintain CR. or sCR, until PD.
Population: Intent-to-treat (ITT) analysis set included all participants who were randomly assigned to the pomalidomide, dexamethasone (Pd) or daratumumab, pomalidomide, dexamethasone (DPd) group.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
percentage of participants | 14.57 [9.36 to 21.22] | 1.96 [0.41 to 5.62]

4. Secondary Outcome: Duration of Response
Description: Duration of response will be restricted to the randomized subjects who achieve a best objective response of PR or better. It is measured from the time, in months, that the criteria for objective response are first met until the date of a progression event (according to the primary definition of PFS).
Time Frame: From informed consent until 30 days after last study treatment, assessed up to approximately 3 years.
Population: Subjects achieving a best objective response of PR or better from the intention-to-treat population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 104 | 71
months | NA [15.21 to NA] — Median and upper limit of 95% CI was not estimable due to short follow-up by participants". | 15.90 [8.31 to 24.80]

5. Secondary Outcome: Time to Next Therapy
Description: Time to next therapy will be defined as the time, in months, from randomization to the date to next anti-neoplastic therapy or death from any cause, whichever comes first.
Time Frame: From randomization until the date to next anti-neoplastic therapy or death from any cause, whichever comes first (approximately up to 3 years)
Population: Intent-to-treat (ITT) analysis set: total of 304 randomized subjects (151 in the Daratumumab/Pomalidomide/Dexamethasone group and 153 in the Pomalidomide/Dexamethasone group).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
months | 23.23 [13.80 to NA] — Upper limit of 95% CI was not estimable due to short follow-up by participants | 11.83 [8.87 to 15.38]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time, in months, from randomization to the date of death from any cause.
Time Frame: From randomization until death from any cause (up to 5 years)
Population: Final OS analysis with the CCO of 31 May 2022 and a median (range) follow-up of 39.6 (0.1-56.9) months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
months | 34.40 [23.69 to 40.25] | 23.72 [19.61 to 29.37]

7. Secondary Outcome: Health-related Quality of Life-Time to Worsening in EORTC QLQ-C30 Scale Scores
Description: Worsening is defined as a decrease in score that is at least half of standard deviation from baseline values, where standard deviation is calculated from the scores at baseline combining both treatment groups.
Time Frame: Approximately up to 3 years (assessed on Day 1 of each treatment cycle, at the end of treatment, and every 4 weeks post treatment until PD.
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
months | 4.01 [2.20 to 7.59] | 3.84 [3.02 to 5.91]

8. Secondary Outcome: Health-related Quality of Life-Time to Worsening in EQ-5D-5L Utility Score
Description: Worsening is defined as a decrease in score that is at least half of standard deviation from baseline values, where standard deviation is calculated from the scores at baseline combining both treatment groups.
  The EQ-5D-5L is a 5 item questionnaire that assesses 5 domains including mobility, self care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today"
Time Frame: Approximately up to 3 years (assessed on Day 1 of each treatment cycle, at the end of treatment, and every 4 weeks post treatment until PD).
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
months | 7.39 [5.32 to 19.52] | 6.14 [3.88 to 13.14]

9. Secondary Outcome: Health-related Quality of Life-Time to Worsening in EQ-5D-5L Visual Analogue Scale
Description: as for outcome 8
Time Frame: as for outcome 8
Population: Intent-to-treat (ITT) analysis set: a total of 304 randomized subjects (151 in the Daratumumab/Pomalidomide/Dexamethasone group and 153 in the Pomalidomide/Dexamethasone group).
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Daratumumab+Pomalidomide+Dexamethasone | Pomalidomide + Dexamethasone
Number analyzed (Participants) | 151 | 153
months | 3.78 [2.83 to 6.54] | 2.86 [1.94 to 3.71]

ADVERSE EVENTS:
Time Frame: Over a median follow-up of 39.6 months (clinical cutoff date: 31 May 2022; approximately an additional 23 months since the primary analysis).
Description: Safety results are summarized for 299 patients (Pd arm: 150; DPd arm: 149).
  Almost all patients in the DPd arm (142/149) received daratumumab SC, per Amendment 1. Of the remaining 7 patients, 4 were switched to daratumumab SC and 3 discontinued treatment before the study was amended to SC administration. The safety information for the DPd arm is presented for all patients who received daratumumab IV and/or SC (n=149) and for patients who received daratumumab SC only (n=142).
Groups:
- Pomalidomide+Dexamethasone: Patients (n=150) received pomalidomide 4 mg orally on Days 1 through 21 of each 28-day treatment cycle and dexamethasone 40 mg (or 20 mg for patients ≥75 years of age) orally on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
- Daratumumab+Pomalidomide+Dexamethasone: Patients (n=149) received: daratumumab SC (fixed dose of 1800 mg) or IV (16 mg/kg) at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, and every 4 weeks (Q4W) thereafter; pomalidomide at a dose of 4 mg orally on Days 1 through 21 of each 28-day treatment cycle; and dexamethasone at a dose of 40 mg (or 20 mg for patients ≥75 years of age) orally on Days 1, 8, 15, and 22 of each 28-day treatment cycle.Only 7 patients received Dara IV and are included in the overall reporting category(DaraPomDex) and the DaraSC subcategory is presented separately to define the safety of the SC dosing regimen.
- Daratumumab (SC)+Pomalidomide+Dexamethasone: Patients (n=142) received: daratumumab SC (fixed dose of 1800 mg) at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, and every 4 weeks (Q4W) thereafter; pomalidomide at a dose of 4 mg orally on Days 1 through 21 of each 28-day treatment cycle; and dexamethasone at a dose of 40 mg (or 20 mg for patients ≥75 years of age) orally on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
- Daratumumab (IV)+Pomalidomide+Dexamethasone: Patients (n=7) received: daratumumab IV (fixed dose of 1800 mg) at weekly intervals (QW) for 8 weeks, then every 2 weeks (Q2W) for an additional 16 weeks, and every 4 weeks (Q4W) thereafter; pomalidomide at a dose of 4 mg orally on Days 1 through 21 of each 28-day treatment cycle; and dexamethasone at a dose of 40 mg (or 20 mg for patients ≥75 years of age) orally on Days 1, 8, 15, and 22 of each 28-day treatment cycle.
Arm/Group | Pomalidomide+Dexamethasone | Daratumumab+Pomalidomide+Dexamethasone | Daratumumab (SC)+Pomalidomide+Dexamethasone | Daratumumab (IV)+Pomalidomide+Dexamethasone
All-Cause Mortality (participants affected / at risk) | 88/150 | 82/149 | 77/142 | 5/7
Serious Adverse Events (participants affected / at risk) | 60/150 | 80/149 | 77/142 | 3/7
Other Adverse Events (participants affected / at risk) | 144/150 | 144/149 | 137/142 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide+Dexamethasone (N=150) | Daratumumab+Pomalidomide+Dexamethasone (N=149) | Daratumumab (SC)+Pomalidomide+Dexamethasone (N=142) | Daratumumab (IV)+Pomalidomide+Dexamethasone (N=7)
Pneumonia (Infections and infestations) | 13 | 23 | 23 | 0 — Pd: 2 deaths DPd: 3 deaths DPd (SC): 3 deaths
Lower respiratory tract infection (Infections and infestations) | 14 | 18 | 18 | 0 — Pd: 1 death DPd: 1 death DPd (SC): 1 death
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 3 | 0
Bronchitis (Infections and infestations) | 5 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 5 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 4 | 4 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 1 — Pd: 0 deaths DPd: 1 death DPd (SC): 0 deaths
Pyrexia (General disorders) | 2 | 3 | 3 | 0
General physical health deterioration (General disorders) | 3 | 1 | 1 | 0
Syncope (Nervous system disorders) | 0 | 4 | 4 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 3 | 3 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 1 | 0 — All deaths are reported as footnotes. The table only refers to the most common SAEs reported with ≥2% higher frequency in the DPd group compared to the Pd group. Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
COVID-19 (Infections and infestations) | 1 | 7 | 7 | 0 — Pd: 1 death DPd: 2 deaths DPd (SC): 2 deaths
Sepsis (Infections and infestations) | 0 | 1 | 1 | 0 — Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
Septic shock (Infections and infestations) | 2 | 1 | 0 | 1 — Pd: 2 deaths DPd: 1 death DPd (SC): 0 deaths
Systemic candida (Infections and infestations) | 0 | 1 | 1 | 0 — Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 — Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 — Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 — Pd: 1 death DPd: 1 death DPd (SC): 1 death
Sudden death (General disorders) | 0 | 1 | 1 | 0 — Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 — Pd: 1 death DPd: 0 deaths DPd (SC): 0 deaths
Hypertensive hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 — Pd: 1 death DPd: 0 deaths DPd (SC): 0 deaths
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 1 | 0 — Pd: 1 death DPd: 0 deaths DPd (SC): 0 deaths
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 — Pd: 1 death DPd: 0 deaths DPd (SC): 0 deaths
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 — Pd: 0 deaths DPd: 1 death DPd (SC): 1 death
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 — Pd: 2 deaths DPd: 0 deaths DPd (SC): 0 deaths
Atypical pneumonia (Infections and infestations) | 1 | 1 | 1 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 1 | 0
Septic shock (Infections and infestations) | 2 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pomalidomide+Dexamethasone (N=150) | Daratumumab+Pomalidomide+Dexamethasone (N=149) | Daratumumab (SC)+Pomalidomide+Dexamethasone (N=142) | Daratumumab (IV)+Pomalidomide+Dexamethasone (N=7)
Neutropenia (Blood and lymphatic system disorders) | 80 | 107 | 103 | 4
Anaemia (Blood and lymphatic system disorders) | 67 | 57 | 55 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 51 | 49 | 48 | 1
Leukopenia (Blood and lymphatic system disorders) | 18 | 39 | 38 | 1
Lymphopenia (Blood and lymphatic system disorders) | 12 | 22 | 19 | 3
Upper respiratory tract infection (Infections and infestations) | 23 | 34 | 31 | 3
Pneumonia (Infections and infestations) | 10 | 11 | 11 | 0
Lower respiratory tract infection (Infections and infestations) | 11 | 20 | 19 | 1
Bronchitis (Infections and infestations) | 16 | 21 | 21 | 0
Fatigue (General disorders) | 37 | 43 | 39 | 4
Asthenia (General disorders) | 25 | 33 | 33 | 0
Pyrexia (General disorders) | 25 | 28 | 27 | 1
Oedema peripheral (General disorders) | 14 | 25 | 24 | 1
Diarrhoea (Gastrointestinal disorders) | 22 | 36 | 35 | 1
Constipation (Gastrointestinal disorders) | 22 | 21 | 21 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 18 | 18 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 20 | 17 | 17 | 0
Tremor (Nervous system disorders) | 14 | 15 | 14 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 20 | 17 | 15 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 18 | 18 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 12 | 16 | 16 | 0
Insomnia (Psychiatric disorders) | 18 | 13 | 12 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 9 | 8 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 15 | 14 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 11 | 19 | 17 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-04): https://cdn.clinicaltrials.gov/large-docs/36/NCT03180736/Prot_SAP_001.pdf